CLINICAL TRIAL: NCT04058392
Title: FULL TITLE: Camu Camu Effects on Circulating LPS and Systemic Immune Activation in ART-treated Participants: the Camu Camu Pilot Study
Brief Title: Camu Camu in ART-treated People Living with HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Jean-Pierre Routy, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTNPT 032
Record Dates: First submitted 2019-05-06; First posted 2019-08-15 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Camu Camu (Experimental): Assessments will be done at baseline, during and after 12 weeks of Camu Camu intake.
  Interventions: Biological: Camu Camu Capsules

INTERVENTIONS:
Biological: Camu Camu Capsules — Camu Camu powder encapsulated (500mg each). 2 capsules per day will be used for this study

SUMMARY:
Persons living with HIV and receiving antiretroviral therapy (ART) remain with inflammation leading to higher risks of cardiovascular diseases, fatty liver and cancer. It has been observed in colitis and in HIV infection that abnormal composition of the gut microbes and leaky gut induce inflammation contributing to diabetes, fatty liver and cardiovascular risks. Abundance of Akkermansia muciniphila in stool, a type of good bacteria acting as a shield on the gut barrier has been shown to prevent obesity, diabetes and to improve cancer treatment response. Health food (prebiotic) increases the frequency of A. muciniphila in overweight individuals.

Dr Marette, a study collaborator from Laval University, has recently published (Gut, 2018) that an extract from a Brazilian fruit called Camu Camu (CC) protects mice from obesity, reduce LPS, a marker for passage of microbes from the gut into the blood and decreases inflammation in association with the frequency of A. muciniphila in stools. The extract of CC is sold in nutritional stores to regulate body fat.

The investigators will invite 22 participants to take 2 capsules of CC daily for 12 weeks in addition to their ART. CC tolerance and changes in blood and stools for inflammation and microbe composition will be evalutated at the end of the 12-week treatment and 8 weeks post-intake. An optional sub study will assess the changes of gut barrier by doing biopsies by colonoscopy.

CC is expected to beassociated with an enrichment of A. muciniphila in stools, combined with reduced gut damage and inflammation.

ELIGIBILITY:
3.2 Inclusion Criteria

Participants will be eligible for the study if they meet the following criteria:

1. Male or female adults ≥18 years of age.
2. Documented HIV-1 infection by Western Blot, Enzyme Immuno Assay (EIA) or viral load assay.
3. On any ART for at least 2 years, with viremia less than 50 copies/ml during the last two years (occasional blips allowed).
4. On a stable ART regimen (same prescription) for at least 3 months.
5. CD4 count >200 and a CD4/CD8 ratio <1 suggesting an increase in inflammation and risk for non-AIDS events.
6. Able to communicate adequately in either French or English.
7. Able and willing to provide written informed consent prior to screening.
8. Women of childbearing potential must have a negative serum pregnancy test.
9. Women of childbearing potential must agree to use one of the following approved methods of birth control while in the study and until 2 weeks after completion:

   1. Complete abstinence from penile-vaginal intercourse from the screening period until two weeks after the study completion.
   2. Double barrier methods (acceptable barrier methods include diaphragm, coil, contraceptive foam, sponge with spermicide, condom); or
   3. Oral, injectable or implant contraceptives plus one barrier method;
   4. Intrauterine device (IUD) plus one barrier method; or
   5. Male partner sterilization confirmed prior to the female participant's entry into the study; this male is the sole partner for that participant.
   6. Approved hormonal contraception, started at least 30 days before screening.
   7. Another method approved by the trial physician with published data showing that the expected failure rate is <1% per year preferably with condom.

   Any contraception method must be used consistently, in accordance with the approved product label, and for the duration of the study until two weeks after study completion.
10. Women of non-child-bearing potential as defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy.
11. Sexually active men with a female partner of childbearing potential must agree to one of the following methods of birth control:

    1. The use at least one barrier method of contraception (e.g. condom) with a female partner using a second approved method of contraception (IUD, hormonal contraceptive pill, diaphragm, spermicide etc.) during the study and until two weeks after study completion.
    2. Be confirmed sterile.
    3. Have had a successful vasectomy.

Exclusion Criteria

Participants are not eligible to participate in the study if they meet any of the following conditions:

1. Known allergy/hypersensitivity to Camu Camu.
2. Current AIDS-related event or serious health condition including systemic infections in the last 3 months.
3. Severe systemic diseases (e.g. uncontrolled hypertension, chronic renal failure), or active uncontrolled infections.
4. Co-infection with active Hepatitis B or C Virus.
5. Current use or have used in the past 3 months: immune-modulatory agents/chemotherapeutics, prophylactic antibiotics35/antibiotics, proton pump inhibitors, phosphate binders, Metformin or Morphine as these drugs can interact with vitamin C or modulate gut microbiota.
6. Diagnosis of diabetes mellitus (HbA1c≥6.5%) as defined by the Canadian Clinical Practice Guidelines for the Prevention and Management of Diabetes42.
7. Frequent use of polyphenol-rich prebiotics (e.g. cranberry and CC powders and/or capsules) in the last 12 months.
8. Statin or other anti-cholesterol treatment use in the last 3 months.
9. Recent changes in dietary habits, intermittent fasting, chronic constipation or laxative use as these can affect gut microbiota.
10. Psychiatric or cognitive disturbance or any illness that could preclude compliance with the study.
11. Current participation in an experimental therapy study or receipt of experimental therapy within the last 6 months.
12. Women who are pregnant, planning to become pregnant, or breast-feeding.
13. A score of higher than 8 on a Full AUDIT questionnaire (See Appendix 1) at the screening visit, suggesting an alcohol abuse problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Reduction of the plasma marker of microbial translocation LPS, assessed using ELISA. | 12 weeks

SECONDARY OUTCOMES:
Safety and tolerability of CC | 20 weeks
  measured by evaluating adverse events, hematology, and serum chemistries over the course of the study. These evaluations will include HIV viral load, glucose levels, a lipid profile and plasma levels of hsCRP and D-dimer.
Changes in gut integrity markers I-FABP, and sST2, measured by ELISA | 12 weeks and 20 weeks
Changes in microbial translocation marker 1-3-b-D-Glucan assessed using the Fungitell assay | 12 weeks and 20 weeks.
Changes in pro-inflammatory markers (IL-1β, IL-6, IL-8, IL-18. IP-10, IL-17A and F, IL-22, and soluble CD14) and anti-inflammatory markers (IL-10) assessed by ELISA. | 12 weeks and 20 weeks
Changes in T-cell and monocyte activation levels assessed by flow cytometry using markers CD38, HLA-DR and PD-1 | 12 weeks and 20 weeks
Changes in A. muciniphila levels in stools using qPCR | 12 weeks and 20 wekks
Changes in microbiota composition and diversity in stools assessed using 16s rDNA sequencing | 12 weeks and 20 wekks
Changes in HIV reservoir size in blood assessed by PCR | 12 weeks and 20 wekks
Evaluate intra-patient variability using data from two baseline visits, approximately two weeks apart from each other to confirm reliability of baseline results. | 2 weeks
Changes in gut mucosa architecture in a subset of participants who will consent to have colon biopsies before and at the end of the 12 weeks of CC treatment. | 12 weeks
Changes in inflammation in gut mucosa biopsy assessed by myeloperoxidase staining before and at the end of the 12 weeks of CC treatment | 12 weeks
Changes in HIV reservoir size in biopsies using qPCR | 12 weeks
Association between baseline gut microbiota composition (16S rDNA sequencing), and markers of gut integrity (I-FABP, tissue staining) and inflammation (T-cell activation, inflammatory cytokines). | 2 weeks

OTHER OUTCOMES:
Exploratory: Difference in HIV reservoir size from Baseline (Visit 0) to 12 weeks post-CC treatment by TILDA, performed on blood samples | 12 weeks
Exploratory: Changes in other markers of gut damage (including plasma REG3α (45)), microbial translocation (such as plasma 16S rDNA) and immune activation (T-cell activation, cytokines) in the blood and gut biopsies. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Routy, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Mcgill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anhe FF, Nachbar RT, Varin TV, Trottier J, Dudonne S, Le Barz M, Feutry P, Pilon G, Barbier O, Desjardins Y, Roy D, Marette A. Treatment with camu camu (Myrciaria dubia) prevents obesity by altering the gut microbiota and increasing energy expenditure in diet-induced obese mice. Gut. 2019 Mar;68(3):453-464. doi: 10.1136/gutjnl-2017-315565. Epub 2018 Jul 31. PMID 30064988
- [Background] Brenchley JM, Price DA, Schacker TW, Asher TE, Silvestri G, Rao S, Kazzaz Z, Bornstein E, Lambotte O, Altmann D, Blazar BR, Rodriguez B, Teixeira-Johnson L, Landay A, Martin JN, Hecht FM, Picker LJ, Lederman MM, Deeks SG, Douek DC. Microbial translocation is a cause of systemic immune activation in chronic HIV infection. Nat Med. 2006 Dec;12(12):1365-71. doi: 10.1038/nm1511. Epub 2006 Nov 19. PMID 17115046
- [Background] Mehraj V, Jenabian MA, Ponte R, Lebouche B, Costiniuk C, Thomas R, Baril JG, LeBlanc R, Cox J, Tremblay C, Routy JP; Montreal Primary HIV Infection, the Canadian Long-Term Non-Progressors Study Groups. The plasma levels of soluble ST2 as a marker of gut mucosal damage in early HIV infection. AIDS. 2016 Jun 19;30(10):1617-27. doi: 10.1097/QAD.0000000000001105. PMID 27045377
- [Background] Jenabian MA, El-Far M, Vyboh K, Kema I, Costiniuk CT, Thomas R, Baril JG, LeBlanc R, Kanagaratham C, Radzioch D, Allam O, Ahmad A, Lebouche B, Tremblay C, Ancuta P, Routy JP; Montreal Primary infection and Slow Progressor Study Groups. Immunosuppressive Tryptophan Catabolism and Gut Mucosal Dysfunction Following Early HIV Infection. J Infect Dis. 2015 Aug 1;212(3):355-66. doi: 10.1093/infdis/jiv037. Epub 2015 Jan 23. PMID 25616404
- [Derived] Isnard S, Fombuena B, Ouyang J, Royston L, Lin J, Bu S, Sheehan N, Lakatos PL, Bessissow T, Chomont N, Klein M, Lebouche B, Costiniuk CT, Routy B, Marette A, Routy JP; Camu Camu Study Group. Camu Camu effects on microbial translocation and systemic immune activation in ART-treated people living with HIV: protocol of the single-arm non-randomised Camu Camu prebiotic pilot study (CIHR/CTN PT032). BMJ Open. 2022 Jan 17;12(1):e053081. doi: 10.1136/bmjopen-2021-053081. PMID 35039291